CLINICAL TRIAL: NCT01164995
Title: Phase II Pharmacological Study With Wee-1 Inhibitor MK-1775 Combined With Carboplatin in Patients With p53 Mutated Epithelial Ovarian Cancer and Early Relapse (< 3 Months) or Progression During Standard First Line Treatment With an Additional Safety and Preliminary Anti-tumor Activity Cohort of Wee-1 Inhibitor AZD1775 Combined With Carboplatin in Patients With Platinum Resistant TP53 Mutated Epithelial Ovarian Cancer
Brief Title: Study With Wee-1 Inhibitor AZD1775 (MK-1775) and Carboplatin to Treat p53 Mutated Refractory and Resistant Ovarian Cancer
Acronym: M10MKO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marloes van Dijk, PhD, The Netherlands Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10MKO / MK1775-009
Record Dates: First submitted 2010-07-09; First posted 2010-07-19 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Epithelial Ovarian Cancer
Keywords: MK-1775; Carboplatin; epithelial ovarian cancer; p53
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — adavosertib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-1775 and carboplatin (Experimental): MK-1775: oral capsules. Carboplatin: intravenous infusion in 30 minutes
  Interventions: Drug: MK-1775 and carboplatin

INTERVENTIONS:
Drug: MK-1775 and carboplatin — Carboplatin will be administered in a dose resulting in AUC5 (i.v. 30 min) at day 1 of each cycle. Concomittantly with the start of the carboplatin infusion 225 mg of MK-1775 will be administered as an oral capsule, followed by 4 additional doses at 12 hour increments ( = 5 BID doses of MK-1775 in 2.5 days in total). One cycle will last 21 days.
  Other Names: CBDCA

SUMMARY:
The purpose of this study is to determine if patients with p53 mutated epithelial ovarian cancer that have been treated with first line treatment (paclitaxel - carboplatin combination therapy) and that have shown early relapse (within 3 months) or progression during treatment will benefit from treatment with Wee-1 inhibitor MK-1775 and carboplatin.

Additional safety and preliminary anti-tumor activity cohort (first patient in 2017):

To determine the safety and preliminary anti-tumor activity (RECIST 1.1) of AZD1775 in combination with carboplatin in platinum resistant p53 mutated epithelial ovarian cancer (relapse within 6 months), NSCLC, SCLC, cervical, and endometrial cancer, in a 21 day schedule.

DETAILED DESCRIPTION:
Platinum-based drugs are used in first line treatment of epithelial ovarian cancer. Despite high overall initial response rates, resistance or early relapse can occur. MK-1775 is a potent and selective inhibitor of Wee-1 kinase, a kinase that regulates the G2/M checkpoint. Since most human cancers retain p53-related G1 checkpoint abnormalities, they are dependent on the G2 checkpoint. Annulment of the G2 checkpoint may therefore make p53 deficient tumor cells more susceptible to anti-cancer agents. The Phase I study with MK-1775 combined with gemcitabine, carboplatin or cisplatin in patients with advanced solid tumors already confirmed target engagement of MK-1775.

In this study Carboplatin will be administered in combination with MK-1775 in a 21 day cycle. Ovarian cancer patients with a p53 mutation based on PCR/sequencing will be eligible for the study. p53 immunohistochemistry (IHC) wil also be performed.

This study is a proof of concept (POC) study. To proof the hypothesis that MK-1775 is more effective in tumors harboring p53 mutations a single stage study with 21 patients will be performed. The final conclusion will then be made as follows: Applying a A'Hern's Single Stage Phase II Design, a minimum of 6 responses (RECIST 1.0 or CA125) out of 21 patients will provide a 61% power to declare an efficacy of at least a 30% (α=0.05). A response of 13% or less would definitively indicate no efficacy of interest.

Patients will remain on treatment until they no longer have clinical benefit from treatment or when toxicity leads to patient withdrawal. Patients will be followed for at least 30 days following their last dose of study therapy, or until death, whichever comes first.

For patients with stable disease follow-up will take place at least until disease progression has been documented = until time of progression. Patients discontinued from the study for unacceptable adverse experiences will be followed until time of progression and until the resolution or stabilization of the adverse experience. These patients with stable disease at the end of treatment or who discontinued for unacceptable adverse experiences will be evaluated every 2 months at the outpatient department, and CA-125 will be determined. In case of CA-125 increase a CT scan will be performed. In patients for whom CA-125 is not a good marker, a CT-scan will need to be performed every 2 cycles (42 days), until disease progression.

In the additional safety and preliminary anti-tumor activity cohort a minimum of 10 patients will be recruited per tumor type. If no partial responses have been documented in a defined tumor type that tumor type will be closed for further recruitment. If at least one patient shows a PR recruitment may continue until 29 (evaluable) patients have been included per tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of epithelial ovarian cancer, and proven p53 mutated pathway by PCR/Sequencing. IHC will also be performed. In the additional safety and efficacy cohort also inclusion of NSCLC, SCLC, cervical and endometrial cancer (only ovarian cancer cohort is pursued)
* Measurable disease on a CT-scan or elevated Cancer Antigen (CA)-125 levels that can be monitored.
* Patients previously received standard 1st line platinum therapy (combined with paclitaxel) for epithelial ovarian cancer, and showed recurrence on or within 3 months of this treatment (relapse within 6 months in the additional safety and efficacy cohort)
* Able and willing to voluntarily give written informed consent.
* Able and willing to undergo blood sampling for pharmacokinetics and pharmacodynamics.
* Life expectancy ≥ 3 months allowing adequate follow up of toxicity evaluation and anti-tumor activity.
* Minimal acceptable safety laboratory values:

  * Absolute neutrophil count (ANC) of ≥ 1.5 x 109 /L (or 1500/m3).
  * Platelet count of ≥ 100 x 109 /L (or 100,000/mm3).
  * Hemoglobin ≥ 5.6 mmol/L (or 9.1 g/dl).
  * Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 2.5 x ULN, or ALAT and ASAT ≥ 5x ULN in case of liver metastases.
  * Renal function as defined by serum creatinine ≥ 1.5 x ULN or creatinine clearance ≥ 60 ml/min for patients with creatinine levels ≥ 1.5 x ULN (by Cockcroft-Gault formula).
* WHO performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* No radio- or chemotherapy within the last 4 weeks prior to study entry (palliative limited radiation for pain reduction is allowed)
* Able and willing to swallow oral medication.
* Able and willing to receive iv medication.
* Negative pregnancy test (urine/serum) for female patients with childbearing potential.

Exclusion Criteria:

* Symptomatic cerebral or leptomeningeal metastases.
* Current participation or previous participation in a study with an investigational compound, or chemo- and/or radiotherapy within 28 days of receiving first dose of study medication. (Palliative limited radiation for pain reduction is allowed only between day 8 and day 21 of the study, and allowed to a limited area to palliate pain.
* No prior radiation therapy to more than 30% of the bone marrow and patient must have recovered for at least 3 weeks from the hematologic toxicity of prior radiotherapy.
* More than 1 prior cytotoxic chemotherapy regimen in initial trial. In the additional safety and efficacy cohort: more than 2 prior cytotoxic chemotherapy regimens.
* Prior stem cell or bone marrow transplant.
* Unresolved (> grade 1) toxicities of previous chemotherapy, excluding alopecia.
* Known hypersensitivity to the components of the combination study therapy or its analogs.
* Patient has had prescription or non-prescription drugs or other products known to be metabolized by CYP3A4, or to inhibit or induce CYP3A4 that cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 days after the last dose of study medication
* Bowel obstructions or motility disorders that may negatively affect oral drug absorption.
* Patients with known alcoholism, drug addiction and/or a history of psychotic disorders who are not suitable for adequate follow up.
* Women who are pregnant or breast feeding.
* Fertile women who do not agree to use a reliable contraceptive method throughout the study.
* Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients.
* Patients with a known history of hepatitis B or C.
* Neurological disease that may render a patient at increased risk for peripheral or central neurotoxicity.
* Clinical history suggestive for Li Fraumeni syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Number and percentage of Participants with Adverse Events | During treatment with carboplatin and MK-1775 AEs will be recorded up to 30 days after treatment (or until death whatever comes first). Treatment will occur until progressive disease
  Descriptive tables that summarize the number and percentage of patients that experience adverse events as categorized in the NCI CTCAE version 4.0 will be generated for the overall population. Laboratory assessments: screening/day 1, 8, 15 of each cycle, and regular physical examination at the start of each cycle or on indication will be performed and followed until 30 days after the end of study (defined as disease progression or unacceptable toxicity (AEs) or patient withdrawal or patient death) or in case of AEs or Stable disease until time of progression.
Radiological antitumor activity | As long as the patient is treated with carboplatin and MK-1775 radiological assessments will be performed every 2 cycles (42 days) until progressive disease occurs, and evaluated in comparison to the baseline scan
  Radiological assessment (CT scan or MRI) per RECIST 1.1

SECONDARY OUTCOMES:
Pharmacokinetics assessments (not in additional safety and efficacy cohort) | Cycle 1: day 1, 2, 3
  Pharmacokinetic analysis will be performed by using nonlinear mixed effect modeling (NONMEM).
  The pharmacokinetic profile of MK-1775, when given in combination with carboplatin, will be determined in plasma and dry blood on day 1,2,3 of cycle 1. Pharmacokinetics of carboplatin, when given in combination with MK-1775, will be determined in plasma and ultrafiltrates on day 1 of cycle 1.
  Correlations between pharmacokinetic data and toxicity are subsequently analyzed for their significance.
Pharmacodynamic assessments (not in additional safety and efficacy cohort) | Cycle 1: Day 1 (pre-dose) and day 3 and Cycle 2: day 1
  Pharmacodynamic changes induced by MK-1775 in combination with carboplatin, measured as changes in pCDC2, will be determined in surrogate tissue (skin). Skin biopsies will be performed on day 1 of cycle 1 (pre-dose) and on day 3 of cycle 1 within 2 hours of the last intake of MK-1775.
  The relationship of various pharmacokinetic parameters to the pharmacodynamic endpoints will also be explored. Disease response, accompanied by available p53-pathway status, will be descriptively summarized.
In the additional safety and preliminary anti-tumor activity cohort | From day of first treatment cycle until end of study (progression or death whatever comes first), assessed up to 24 months (estimated)
  Progression free survival

OTHER OUTCOMES:
Biomarker analyses in additional safety and efficacy cohort | Biopsies will be obtained before treatment (baseline), on treatment in case of response and at time of progression
  WGS and IHC staining for determination of predictive biomarkers for resistance and response

CONTACTS AND LOCATIONS:
Overall Officials: FL Opdam, MD PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- FL Opdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Embaby A, Kutzera J, Geenen JJ, Pluim D, Hofland I, Sanders J, Lopez-Yurda M, Beijnen JH, Huitema ADR, Witteveen PO, Steeghs N, van Haaften G, van Vugt MATM, de Ridder J, Opdam FL. WEE1 inhibitor adavosertib in combination with carboplatin in advanced TP53 mutated ovarian cancer: A biomarker-enriched phase II study. Gynecol Oncol. 2023 Jul;174:239-246. doi: 10.1016/j.ygyno.2023.05.063. Epub 2023 May 24. PMID 37236033
- [Derived] Leijen S, van Geel RM, Sonke GS, de Jong D, Rosenberg EH, Marchetti S, Pluim D, van Werkhoven E, Rose S, Lee MA, Freshwater T, Beijnen JH, Schellens JH. Phase II Study of WEE1 Inhibitor AZD1775 Plus Carboplatin in Patients With TP53-Mutated Ovarian Cancer Refractory or Resistant to First-Line Therapy Within 3 Months. J Clin Oncol. 2016 Dec 20;34(36):4354-4361. doi: 10.1200/JCO.2016.67.5942. Epub 2016 Oct 28. PMID 27998224